CLINICAL TRIAL: NCT05425992
Title: Improving Communication With and Building a Stronger Medical Home Among Spanish-speaking Families in the Center for Cancer and Blood Disorders
Brief Title: Improving Communication and Building a Stronger Medical Home Among Spanish-speaking Families
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 21-4238.cc; NCI-2022-04061 (Other: CTRP)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Leukemia; Non Hodgkin Lymphoma
Keywords: Spanish-speaking
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated in CCBD: Patients who are currently receiving therapy at the Center for Cancer and Blood Disorders
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patient/parent dyads expressing interest will be interviewed by a bilingual Spanish certified provider via televideo with as needed interpreter support. Interviews will be audio recorded for review and translation purposes and then will be destroyed. Interview format will be supportive and information seeking only with reassurance that purpose is for care improvement and that all answers will be evaluated without association to patient name. Interviews will then be translated and reviewed by the PI for themes regarding perceived clinic successes and perceived clinic barriers in communication or care.

SUMMARY:
This study will seek to improve communication with Spanish speaking families and patients with Cancer and Blood Disorders.

DETAILED DESCRIPTION:
The Principal Investigator seeks to improve communication with Spanish speaking families with the following goals: 1) to increase patient and family sense of inclusion in the medical community, 2) to increase patient and family medical knowledge and understanding, 3) to improve patient adherence with critical medical regimens, and ultimately, 4) to increase equality of comprehensive medical care delivery across the continuum of care including physical and psychosocial domains.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 22 years of age
* Diagnosis of leukemia or non-Hodgkin lymphoma
* Spanish as preferred language for patient, parent or guardian
* Received or receiving care at the Center for Cancer and Blood Disorders (CCBD)

Exclusion Criteria:

* Patients without oncologic diagnosis
* Patients with parents whose language preference is English
* Patients who received care solely outside of the CCBD

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients eligible for enrollment are identified from EPIC electronic medical record with notification for newly diagnosed families of Spanish language preference.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine a baseline level of Spanish speaking patient satisfaction of care | 12 months
  Understand the patient experience using qualitative interview of Spanish speaking patients and families Determine satisfaction based on open-ended question with unsatisfied to satisfied as markers.
Determine a baseline level of Spanish Speaking family satisfaction of care | 12 months
  Understand the patient experience using qualitative interview of Spanish speaking patients and families Determine satisfaction based on open-ended question with unsatisfied to satisfied as markers.
Determine effects of language barrier on Spanish speaking patient needs | 12 months
  Understand the patient experience using qualitative interview of Spanish speaking patients and families.
  Determine satisfaction based on open-ended question to determine a list or pattern of common patient needs.
Determine the effect of language barrier on barriers to patient care | 12 months
  Understand the patient experience using qualitative interview of Spanish speaking patients and families.
  Determine satisfaction based on open-ended question to determine a list or pattern of common barriers to patient care.
Effect of language barrier on efficiency of access to care | 12 months
  Understand the patient experience using qualitative interview of Spanish speaking patients and families.
  Determine satisfaction based on open-ended question to determine how quickly patient was able to receive care.

SECONDARY OUTCOMES:
Determine patient interest in home telemedicine support program | 12 months
  Open-ended questions will be used to determine level of interest in a telemedicine support program.
Determine patient interest in home telemedicine support program after discharge | 12 months
  Open-ended questions will be used to determine level of interest in a telemedicine support program to be used after discharge from hospital.
Determine Spanish speaking patient interest in telemedical check-ins during intensive phases of therapy | 12 months
  Open-ended questions will be used to determine level of interest in a telemedical support during treatment.
Determine Spanish speaking patient interest in medication assistance during intensive phases of therapy | 12 months
  Open-ended questions will be used to determine level of interest in a telemedical medication support during therapy.
Determine Spanish speaking patient interest in medical check-ins during maintenance | 12 months
  Open-ended questions will be used to determine level of interest in a telemedical check-ins during maintenance.
Determine Spanish speaking patient interest in medication assistance during maintenance | 12 months
  Open-ended questions will be used to determine level of interest in a telemedical medication assistance during maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Rogers, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No